CLINICAL TRIAL: NCT07056660
Title: Efficacy and Safety of Atmospheric Pressure Cold Plasma in the Treatment of Moderate-to-severe Tinea Pedis: a Prospective, Randomized, Double-blind, Placebo-controlled Multicenter Clinical Trial
Brief Title: Atmospheric Pressure Cold Plasma for Moderate-to-severe Tinea Pedis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shenyang Medical College (Other)
Collaborators: Tsinghua University (Other)
Responsible Party: Principal Investigator, Lin Tao, MM, Shenyang Medical College
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 630pedis
Record Dates: First submitted 2025-06-30; First posted 2025-07-09 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Tinea Pedis
Keywords: Tinea pedis; Atmospheric pressure cold plasma
MeSH Terms: conditions — Tinea Pedis | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: In the placebo group, the electric field for plasma generation will remain off, so no plasma will be produced; only operational sounds will be simulated to maintain procedural blinding.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CAP group (Active Comparator)
  Interventions: Device: Active CAP therapy; Other: standard care
- Sham group (Placebo Comparator)
  Interventions: Device: Sham CAP therapy; Other: standard care

INTERVENTIONS:
Device: Active CAP therapy — The CAP group will additionally undergo atmospheric pressure cold plasma (CAP) treatment (plasma-activated gas form, CAP-Activated Gas; patent number: ZL202110209052.X, provided by Xi'an Jiaotong University), once daily for the first five days and every other day thereafter, for a total of 13 sessions. Each session will involve enclosing the target area in a treatment bag sealed with medical adhesive tape; plasma-activated gas rich in ozone (O₃) will be delivered and recirculated for 20 minutes, followed by plasma-activated gas rich in nitric oxide (NO) for an additional 5 minutes, in strict accordance with the standard operating procedures provided by the manufacturer.
  Arms: CAP group
Device: Sham CAP therapy — In the placebo group, the electric field for plasma generation will remain off, so no plasma will be produced; only operational sounds will be simulated to maintain procedural blinding.
  Arms: Sham group
Other: standard care — The group will receive standard care according to current clinical guidelines

SUMMARY:
Tinea pedis (athlete's foot) is a common and highly contagious fungal infection of the feet. Moderate-to-severe cases present with extensive skin lesions, severe symptoms, frequent recurrences, and increased risk of complications, often proving refractory to conventional topical therapies. Anatomical niches, poor drug penetration, and antifungal resistance make effective management challenging and negatively impact patients' quality of life.

Current treatments, including topical and systemic antifungals or physical modalities, are often limited by incomplete efficacy, complexity, or poor adherence. Therefore, more effective and practical treatment options are urgently needed.

Atmospheric pressure cold plasma (CAP) is an innovative technology that generates reactive species capable of targeting pathogens while preserving normal tissue. CAP has demonstrated strong antimicrobial effects and promotes wound healing in biomedical research. This study will evaluate the efficacy and safety of CAP in treating moderate-to-severe tinea pedis, aiming to address unmet clinical needs and support future clinical application.

DETAILED DESCRIPTION:
Tinea pedis, commonly known as athlete's foot, is a highly contagious dermatophytic infection of the feet, characterized by erythema, desquamation, vesicles, and sometimes thickening or fissuring of the skin. It remains one of the most prevalent skin diseases worldwide, especially in hot and humid environments, which favor fungal growth and transmission. Typical clinical manifestations include blistering, scaling, and itching between the toes, on the heels, and the lateral aspects of the foot; in severe cases, patients may experience maceration, exudation, and secondary bacterial infections.

Moderate-to-severe tinea pedis is associated with extensive skin involvement, more intense symptoms (such as severe pruritus, pain, and functional impairment), frequent recurrences, and an increased risk of complications including cellulitis and chronic wounds. These forms of the disease are not only more refractory to conventional topical therapies, but also have a significant impact on patients' quality of life and daily functioning. Persistent or extensive lesions are more likely to harbor residual fungi in anatomical niches (e.g., toe webs, heel fissures), leading to repeated treatment failures and contributing to transmission within households and the wider community. Therefore, improving the efficacy of fungal inactivation and reducing recurrence rates in moderate-to-severe tinea pedis is a key unmet need in dermatology.

Over the years, multiple approaches have been explored for superficial fungal eradication, including preventive measures, physical therapies, and chemical agents. However, current treatments face several limitations: (1) the complex anatomical structure and irregular surface of the foot make it difficult for topical agents or sterilization procedures to penetrate all affected areas, often leaving residual fungi; (2) dermatophytes have substantial survival capacity and may develop resistance, making mild or insufficient therapies less effective for complete eradication; (3) many existing treatment modalities are cumbersome, require complex procedures, or lack flexibility, limiting their widespread use and patient adherence. As a result, achieving both effective fungal eradication and practical, patient-friendly treatment options remains an important clinical challenge, especially for moderate-to-severe cases.

Atmospheric pressure cold plasma (CAP) represents an innovative fourth-state physical technology, capable of generating a high density of energetic electrons, ions, excited atoms, and reactive species (including ROS and RNS) at near-room temperature. This technology has been widely adopted for material processing, environmental protection, new energy applications, and increasingly, for biomedical purposes. In medical research, CAP-generated reactive agents, ultraviolet irradiation, and thermal effects have been shown to disrupt microbial cell structures, induce apoptosis, and promote tissue regeneration by stimulating growth factor expression and enhancing wound healing processes. Importantly, CAP offers selective cytotoxicity, enabling targeted inactivation of pathogenic microorganisms while preserving normal tissue viability through adjustable plasma parameters.

Given its potent antimicrobial effects, safety profile, and unique physical-chemical mechanisms, CAP is a highly promising candidate for the treatment of recalcitrant cutaneous infections, such as moderate-to-severe tinea pedis. Applying CAP to the management of tinea pedis could potentially address the unmet needs of deeper fungal eradication, reduced recurrence, and improved patient outcomes, particularly in those with more extensive, symptomatic, or difficult-to-treat disease.

Based on this rationale, the present study will evaluate the efficacy and safety of CAP in the treatment of moderate-to-severe tinea pedis, providing important supporting evidence for larger-scale clinical applications in the future.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 70 years, irrespective of sex.
* Clinical diagnosis of interdigital tinea pedis (non-hyperkeratotic type), with or without extension to other areas, of moderate to severe intensity, defined as follows: target lesion(s) will have an erythema score of ≥2 and either a desquamation or pruritus score of ≥2, with a total score ≥4 (using a 0-3 scale for each item).
* Positive direct potassium hydroxide (KOH) microscopic examination for dermatophytes.
* Women of childbearing potential will agree to use effective contraception throughout the study period.
* Written informed consent will be obtained prior to enrollment.

Exclusion Criteria:

* Severe bacterial infection or other dermatological conditions that may interfere with study assessments.
* Serious cardiac, hepatic, or renal diseases, diabetes mellitus, or major psychiatric disorders.
* Systemic corticosteroid or immunosuppressant use within the past 3 months.
* Systemic antifungal agents within the past 2 months or topical antifungal agents within the past 2 weeks.
* Pregnancy or breastfeeding.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2025-07-25 (Actual); Primary Completion 2026-07-15 (Estimated); Study Completion 2026-08-20 (Estimated)

PRIMARY OUTCOMES:
Change in lesion area | Baseline (V0) and at each visit within 20 ± 1 days after randomization (V1-V13)
  Assessments are conducted daily for the first five days (V1-V5), and every two days thereafter (V6-V13).

SECONDARY OUTCOMES:
Time to 10% reduction in lesion area | Assessment time points: Baseline (V0) and at each visit within 20 ± 1 days after randomization (V1-V13).
Change in quality of life as measured by the EQ-5D questionnaire | Baseline and at the last visit during the treatment period (V1, V13).
Change in quality of life as measured by the SF-12 questionnaire | Baseline and at the last visit during the treatment period (V1, V13).
Incidence of skin irritation | Baseline (V0) and at each visit within 20 ± 1 days after randomization (V1-V13).
Incidence of local burning sensation | Baseline (V0) and at each visit within 20 ± 1 days after randomization (V1-V13).

OTHER OUTCOMES:
Change in quality of life as measured by the EQ-5D questionnaire | Baseline and at follow-up visits at 180 ± 15 days and 360 ± 20 days after randomization (V1, V14, V15).
Change in quality of life as measured by the SF-12 questionnaire | Baseline and at follow-up visits at 180 ± 15 days and 360 ± 20 days after randomization (V1, V14, V15).

CONTACTS AND LOCATIONS:
Overall Officials: Yun-En Liu, MD, Study Chair — Shenyang Medical College; Lin Tao, MM, Principal Investigator — Shenyang Medical College
Locations (1):
- The 989th Hospital of Chinese People's Liberation Army Joint Logistic Support Force, Luoyang, Henan, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol